CLINICAL TRIAL: NCT00697957
Title: Bone Adaptation to Impact Loading - Significance of Loading Intensity
Brief Title: Bone Adaptation to Impact Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu Deaconess Institute (Other); UKK Institute (Other); Finnish Institute of Occupational Health (Other); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government); Newtest Ltd (Unknown); CCC Group Ltd. (Industry); Fastrax Ltd. (Industry)
Responsible Party: Timo Jämsä, professor, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 40093/02
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Osteoporosis
Keywords: acceleration; bone density; cardiovascular diseases; exercise; female; fragility fractures; impact intensity; intervention studies; osteoporosis; premenopause
MeSH Terms: conditions — Osteoporosis; Cardiovascular Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): Control group
- 1 (Experimental): Exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Progressive impact exercise
  Arms: 1

SUMMARY:
Ageing populations have made osteoporosis and fragility fractures a major public health concern worldwide. Half of all women and 30% of all men will suffer a fracture related to osteoporosis during their lifetime. While medical prevention of this immense problem is impossible at population level, it is necessary to find efficient preventive strategies. Exercise is one of the major prevention approaches because one reason behind the increasing burden of osteoporosis is the modern sedentary lifestyle. However, the optimal type, intensity, frequency, and duration of exercise that best enhances skeletal integrity are still largely unknown.

We conducted a 12-month population-based randomized controlled exercise intervention in 120 premenopausal women. The aim was to investigate the effect of impact exercise on bone mineral density, geometry and metabolism in healthy women with the intention of assessing the intensity and amount of impact loading with a novel accelerometer-based measurement device. Training effects on risk factors of osteoporotic fractures, physical performance and risk factors of cardiovascular diseases were also evaluated.

This study demonstrated that 12 months of regular impact exercise favoured bone formation, increased bone mineral density in weight-bearing bones, especially at the hip, and led to geometric adaptations by increasing periosteal circumference. Bone adaptations had a dose- and intensity-dependent relationship with measured impact loading. Changes in proximal femur were threshold-dependent, indicating the importance of high impacts exceeding acceleration of 4 g as an osteogenic stimulus. The number of impacts needed to achieve this stimulation was 60 per day. Impact exercise also had a favourable effect on physical performance and cardiorespiratory risk factors by increasing maximal oxygen uptake, dynamic leg strength and decreasing low-density lipoproteins and waist circumference. Changes were dose-dependent with impact loading at wide intensity range.

Bone adapts to impact loading through various mechanisms to ensure optimal bone strength. The number of impacts needed to achieve bone stimulation appeared to be 60 per day, comparable to the same number of daily jumps. If done on a regular basis, impact exercise may be an efficient and safe way of preventing osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Random population-based sample of women:

  * Age 35-40 yr
  * residing in the city of Oulu, Finland
  * in March 2002

Exclusion Criteria:

* cardiovascular, musculoskeletal, respiratory, or other chronic diseases that might limit training and testing
* diseases or medication affecting the bone
* pregnancy and breastfeeding
* regular current or previous participation in impact-type exercises and long-distance running more than three times a week

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2002-05; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
bone mineral density | 0 and 12 months

SECONDARY OUTCOMES:
muscle strength | 0 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oulu, Oulu, Finland

REFERENCES:
- [Derived] Ahola R, Korpelainen R, Vainionpaa A, Leppaluoto J, Jamsa T. Time-course of exercise and its association with 12-month bone changes. BMC Musculoskelet Disord. 2009 Nov 12;10:138. doi: 10.1186/1471-2474-10-138. PMID 19909496